CLINICAL TRIAL: NCT03084926
Title: A Phase 1, First-in-human, Single-arm, Multi-center, Open-label, Repeated-Dose, Dose-escalation Study to Assess Safety, Tolerability and Pharmacokinetics of MP0274 in Patients With Advanced HER2-positive Solid Tumors
Brief Title: First-in-human Study to Investigate Safety, Blood Levels and Activity of MP0274 in Cancer Patients With HER2-positive Solid Tumors
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Molecular Partners AG (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MP0274-CP101; 2016-004712-36 (EudraCT Number)
Record Dates: First submitted 2017-03-06; First posted 2017-03-21 (Actual); Last update posted 2022-01-10 (Actual); Status verified 2022-01

CONDITIONS: Neoplasms
MeSH Terms: conditions — Neoplasms

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- MP0274 (Experimental)
  Interventions: Drug: MP0274

INTERVENTIONS:
Drug: MP0274 — Intravenous infusion of MP0274 as single agent at four planned dose levels, every three weeks until progressive disease, unacceptable toxicity or patient withdrawal for other reasons

SUMMARY:
This study is investigating a new experimental therapy, MP0274, a DARPin® drug candidate targeting HER2. Preclinical studies suggest that MP0274 may provide additional benefit for the treatment of HER2-positive cancers. This is the first study of MP0274 in humans and its main purpose is to test its safety and tolerability in patients with HER2-positive cancer. This study will also examine the blood levels of MP0274 at several escalating dose levels and a recommended dose for further development will be determined. The recommended dose will be tested in a second part of the study to confirm safety and to further assess the preliminary biologic and anti-tumor activity

ELIGIBILITY:
INCLUSION CRITERIA

1. Have signed and dated written informed consent prior to performing any study procedure, including screening
2. Are ≥ 18 years old on the day of signing informed consent
3. Have histologically confirmed and documented HER2 positive solid tumor malignancy that is unresectable, locally advanced, or metastatic with progression

   * Part A of study: Assessed on tumor tissue from most recent biopsy
   * Part B of study: Assessed on the latest tumor biopsy material for HER2 and other scheduled tissue testing from within 6 months before entry into the study Part A and B: Tumor tissue must be made available to the Sponsor for central testing
4. Have received standard, available therapies approved for their cancer, unless they are unsuitable for these treatments (incurable disease)

   * Have documented PD on most recent systemic antitumor treatment
   * Disease assessment Part A: Evaluable Disease (disease that cannot be measured directly by the size of the tumor but can be evaluated by other methods) or Measurable Disease according to RECIST v1.1 (in case of skin lesions, documentation by color photography including a ruler to estimate the size of the lesion is acceptable) Part B: Measurable Disease as per RECIST 1.1
5. Have an ECOG PS of 0-2
6. Have adequate hematological function prior to first scheduled dose, defined as:

   * Absolute neutrophil count ≥ 1500 cells/µL
   * Hemoglobin ≥ 9 g/dL
   * Platelet count ≥ 75,000/µL
   * Prothrombin time or activated partial thromboplastin (aPTT) time ≤ 1.5 × upper limit of normal (ULN)
7. Adequate renal function prior to first scheduled dose, defined as either:

   * Serum creatinine ≤ 1.5 mg/dL Or
   * Serum creatinine clearance ≥ 40 mL/min (by Cockcroft-Gault equation)
8. Values for potassium, calcium and magnesium must be within normal ranges. Patients may receive supplements to meet these requirements
9. Adequate hepatic function

   * Aspartate aminotransferase (AST)/ alanine aminotransferase (ALT) ≤ 2.5 × ULN, or if known hepatic metastases ≤5 × ULN
   * Total bilirubin ≤ 1.5 × ULN
10. Serum albumin concentration ≥ 30 g/L
11. Highly effective contraception, for both women and men, is ensured:

    * Female patients must be either post-menopausal women, or highly effective contraceptive measures must be ensured. Menopause is defined as occurring 12 months after last menstrual period
    * Pre-menopausal or menopausal women who fulfill the following conditions: They must have had a prior hysterectomy or be using 2 highly effective methods of contraception (i.e. with failure rates less than 1% per year when used consistently and correctly, e.g. established use of oral, injected or implanted hormonal methods of contraception; intrauterine device; condom with spermicidal foam or gel or film or cream or suppository), from the time of screening through the whole treatment phase of the study, and for at least 3 months following the completion of the last MP0274 administration
    * Men capable of fathering a child must agree to use barrier contraception (combination of a condom and spermicide) or limit activity to post-menopausal, surgically sterilized, or a contraception-practicing partner, during the treatment phase of the study and for at least 3 months following the completion of the last MP0274 infusion
    * Men capable of fathering a child must refrain from donating sperm for duration of study and for at least 4 months after last administration of MP0274
12. Female patients of child-bearing potential must have a negative serum pregnancy test result at screening

EXCLUSION CRITERIA

Patients will be ineligible if 1 or more of the following statements are applicable:

1. Hematological malignancies or other second primary malignancy, that is currently clinically significant or requires active intervention
2. Known brain metastases that are clinically unstable despite treatment with anticonvulsives and/or corticosteroids for at least 8 weeks prior to first scheduled dose of MP0274
3. Receipt of any of the following previous anti-tumor treatments:

   * Cumulative doxorubicin ≥ 360 mg/m2
   * Cumulative epirubicin ≥ 720 mg/m2
   * Lapatinib within 7 days of scheduled dosing Day 1
   * Chemotherapy, trastuzumab, or trastuzumab emtansine, other biologics, targeted or experimental therapy within 4 weeks of scheduled dosing Day 1, and for pertuzumab within 12 weeks
   * Nitrosoureas or mitomycin C chemotherapy within 6 weeks of scheduled dosing Day 1
   * Hormonal (e.g. tamoxifen) or aromatase inhibitor therapy within 8 weeks prior to first dose MP0274, except if no change in dose or schedule 8 weeks prior to first scheduled dose MP0274
   * Newly initiated therapy with bisphosphonate or receptor activator of nuclear kappa-B ligand (RANKL)-therapy within 8 weeks prior to first scheduled dose MP0274. If stable on dosing schedule for more than 8 weeks prior to first scheduled dose MP0274 these therapies are allowed. However, no new therapy with bisphosphonate/RANKL is allowed during the course of the study
4. Received concurrent radiation therapy within 4 weeks prior to first scheduled dose MP0274. Local radiation therapy to painful bone metastases following institutional standard practice for palliative radiotherapy to bone metastases is allowed
5. Presence of neuropathy as residual toxicity after prior anti-tumor therapy Grade > 2
6. Any of the following cardiac exclusion criteria:

   * Known history of symptomatic congestive heart failure
   * LVEF < 55%, assessed by 2-dimensional echocardiography (2D Echo)
   * Known absolute decrease in LVEF of ≥ 15 absolute percentage points on prior anti-HER2 therapy, even if asymptomatic
   * High-risk uncontrolled arrhythmias such as resting bradycardia with a heart rate < 55 beat/min, atrial tachycardia with a resting heart rate > 100 beats/min, clinically significant ventricular arrhythmia (ventricular tachycardia) or higher-grade atrioventricular (AV) block (second degree AV-block Type 2 or third degree AV-block), implantable pacemaker or defibrillator, family history of long QT syndrome
   * QTc prolongation > Grade 1 (> 480 ms) at screening measured on 2 separate ECGs at least 10 min apart
   * Angina pectoris requiring anti-angina medication
   * History of cardiac infarction or evidence of transmural infarction on ECG
   * Troponin ≥ Grade 1 (above the upper limit of normal)
   * Both, CK > 2.5-fold ULN range and CK-MB > 6% of total CK at screening
   * Coronary artery bypass graft, coronary artery angioplasty or stent placement within 12 months before screening
   * Clinically significant valvular heart disease
7. Known hyperthyroidism
8. Hypertension which is not controlled to systolic < 160 mm Hg and diastolic < 100 mm Hg
9. Clinically significant lung disorders such as:

   * Non-malignant interstitial lung disease or pneumonitis
   * Dyspnea of any cause requiring supplemental oxygen therapy and dyspnea at rest due to complications of advanced malignancy and co-morbidities
10. History of allogeneic bone marrow or stem cell transplant
11. Known positivity for human immunodeficiency virus (HIV) or history of HIV
12. Patients having active hepatitis B (chronic or acute; defined as having a positive hepatitis B surface antigen [HbsAg] test at screening) or active hepatitis C at screening

    o Patients with past hepatitis B virus (HBV) infection or resolved HBV infection (defined as the presence of hepatitis B core antibody [HbcAb] and absence of HbsAg) are eligible. Patients positive for hepatitis C virus (HCV) antibody are eligible only if polymerase chain reaction is negative for HCV RNA
13. Any active infection requiring the use of parenteral anti-microbial agents or that is > Grade 2
14. Unable or unwilling to comply with all study requirements for clinical visits, examinations, tests, and procedures
15. Concurrent participation in another clinical study involving treatment with the IMP and/or safety follow-up post treatment with IMP (Long-term Survival Follow-up is permitted)
16. Previous treatment with MP0274 (to exclude re-entering the study)
17. Hypersensitivity to any of the excipients of the finished drug MP0274
18. Patients who are pregnant or breast-feeding

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 22 (Actual)
Dates: Start 2017-08-08 (Actual); Primary Completion 2021-12-13 (Actual); Study Completion 2021-12-13 (Actual)

PRIMARY OUTCOMES:
Incidence and severity of adverse events | from first infusion to end-of-study visit, up to 12 months
  Number and grading according to the National Cancer Institute Common Terminology Criteria for Adverse Events (NCI CTCAE)

SECONDARY OUTCOMES:
Pharmacokinetics of MP0274 | from first infusion to end-of-study visit, up to 12 months
  Serum concentration-time profile of MP0274
Preliminary assessment of anti-tumor activity of MP0274 | from first infusion to end-of-study visit, up to 12 months
  Efficacy evaluation based on Response Evaluation Criteria in Solid Tumors (RECIST)
Incidence of anti-drug-antibodies | from first infusion to end-of-study visit, up to 12 months
  Serum concentration-time profile of anti-drug antibodies

CONTACTS AND LOCATIONS:
Locations (4):
- Germany (2):
  - Study Site Frankfurt, Frankfurt
  - Study Site Heidelberg, Heidelberg
- Study Site St. Gallen, Sankt Gallen, Canton of St. Gallen, Switzerland
- Study Site Cambridge, Cambridge, United Kingdom